CLINICAL TRIAL: NCT05613166
Title: A Prospective, Randomized, Double-blind, Placebo-Controlled Phase Ⅱ Study to Evaluate the Efficacy of Adjunctive Everolimus Treatment in Patients With Refractory Epilepsy
Brief Title: Adjunctive Everolimus Treatment of Refractory Epilepsy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute on Drug Dependence, China (Other)
Collaborators: Peking University (Other); Shengjing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PKU-SJ-01-2021-V1
Record Dates: First submitted 2022-11-05; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Epilepsy
Keywords: everolimus
MeSH Terms: conditions — Epilepsy | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- everolimus 1h (Experimental): The study participants will orally receive everolimus within 1 hour and placebo at 8-9 hours after each seizure event, but with intervals longer than 24 hours.
  Interventions: Drug: Everolimus; Drug: Placebo
- everolimus 8-9h (Experimental): The study participants will orally receive placebo within 1 hour and everolimus at 8-9 hours after each seizure event, but with intervals longer than 24 hours.
  Interventions: Drug: Everolimus; Drug: Placebo
- placebo (Placebo Comparator): The study participants will orally receive placebo both within 1 hour and at 8-9 hours after each seizure event, but with intervals longer than 24 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Everolimus — Everolimus will be administrated orally based on seizure events, with an administration interval longer than 24 hours. Participates with a body surface area (BSA) of <= 1.2 m^2, the dosage was 2.5 mg/time; for BSA 1.3-2.1 m^2, the dosage was 5 mg/time; and for BSA >=2.2 m^2, the dosage was 7.5 mg/time.
  Other Names: Afinitor
  Arms: everolimus 1h; everolimus 8-9h
Drug: Placebo — Vitamin C

SUMMARY:
This project is a prospective, randomized, placebo-controlled, double-blind study that will evaluate the clinical efficacy of everolimus as an adjunctive treatment in adult patients diagnosed with refractory epilepsy.

DETAILED DESCRIPTION:
The project consists of a screening and baseline monitoring period of 1-2 weeks, and a treatment period of 1 week, followed by a 3-month follow-up period. Approximately 108 participants will be randomized in a blinded manner to one of three arms in a 1:1:1 fashion (everolimus 1h : everolimus 8-9h : Placebo). After screening, participants will have the first video-EEG monitoring for up to 24 hours to assess baseline levels, followed by 1 week of treatment, the second video-EEG monitoring, and a 3-month post treatment follow-up period. During the treatment period, participants will be given everolimus or placebo directed to seizure events. In the "everolimus 1h" group, everolimus will be administrated immediately after seizure events (within 1 hour); while in the "everolimus 8-9h" group, everolimus administration will be delayed (at 8-9 hours after seizure events). We conduct this study to assess the efficacy of everolimus in adult refractory epilepsy patients under an administration strategy in a limited time window immediately after seizure events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of drug resistant epilepsy, with treatment of at least two approved anti-epileptic drugs (AEDs), and having at least one reported seizure per month during the 3-month baseline phase and no continuous 3-month seizure-free period.
* Diagnosis of focal epilepsy without secondary generalization.
* Treatment with a stable dose of AEDs that must have no drug interactions with everolimus (eg, valproic acid, topiramate, oxazepine, phenobarbital, phenytoin, and primidone) for at least 12 weeks before enrollment.

Exclusion Criteria:

* History of non-drug treatment for epilepsy, eg, vagus nerve stimulation (VNS), ketogenic diet, and epilepsy surgery.
* Severe dysfunction in kidney.
* With significant infectious, immunologic, or oncologic comorbidity at the time of enrollment.
* Currently taking or previously treated systemically with an mammilian target of rapamycin (mTOR) inhibitor.
* History of seizures secondary to drug abuse, psychogenic nonepileptic seizures, or an episode of status epilepticus within 1 year before enrollment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline frequency of epileptic discharge | 1 week
  Comparing frequency of epileptic discharge during video-EEG monitoring after versus before treatment

SECONDARY OUTCOMES:
Change from baseline seizure frequency | 6 months
  Comparing number of seizures in 3 months after treatment versus baseline
Change from baseline seizure types | 6 months
  Comparing types of seizures in 3 months after treatment versus baseline
Change from baseline frequency of seizure-free days | 6 months
  Comparing seizure-free days in 3 months after treatment versus baseline
Seizure-free rate | 3 months
  Patients remaining seizure free in 3 months after treatment
Change from baseline occurrence of secondary generalized seizure and status epilepticus | 6 months
  Comparing number of occurrence of secondary generalized seizure and status epilepticus in 3 months after treatment versus baseline
Quality of life questionnaire (QOLIE-31-Chinese version) scores | 3 months
  Comparing the scores at 3 months after treatment versus before treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China